CLINICAL TRIAL: NCT04322981
Title: Pharmacist-led Hepatitis C Diagnosis and Rapid Management - in Community
Brief Title: Pharmacist-led Hepatitis C Management
Acronym: PHARM-C
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-5265
Record Dates: First submitted 2020-02-20; First posted 2020-03-26 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis C Virus Infection
Keywords: Point-of-care testing; Rapid access to treatment; Pharmacist-led; Service co-localization
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Screening, evaluation and treatment at an outpatient pharmacy compared to referral to hepatology clinics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Pharmacist-Led (Experimental): Patients in Arm 1 will receive care and treatment at their home pharmacy and be evaluated and treated by a community pharmacist under medical directives and with study oversight.
  Interventions: Behavioral: Pharmacist-Led care
- Academic hepatology (Active Comparator): Patients in Arm 2 will be evaluated and treated by hepatologists at the Toronto Centre for Liver Disease.
  Interventions: Behavioral: Standard of Care (Hepatology)

INTERVENTIONS:
Behavioral: Pharmacist-Led care — Rapid testing in a community pharmacy, with rapid linkage to care and treatment that is pharmacist-led
  Arms: Community Pharmacist-Led
Behavioral: Standard of Care (Hepatology) — Rapid testing in a community pharmacy, with standard of care referral to academic hepatology
  Arms: Academic hepatology

SUMMARY:
Hepatitis C virus (HCV) continues to disproportionately affect vulnerable and marginalized persons in Canada. During the interferon treatment era, certain circumstances precluded individuals from receiving treatment, most notably mental health concerns or active substance use. In addition to the tolerability and efficacy of all-oral direct acting antivirals (DAAs), novel diagnostic strategies have also increased engagement in the care cascade. Point-of care and/or dried blood spot antibody as well as RNA testing allow for diagnosis without the need for phlebotomy, a major barrier for those with a history of past or current injection drug use. Despite these advances in diagnostic streamlining and increased cure rates, engagement post-diagnosis continues to be a major gap. Although the exact mechanism of HCV acquisition may not be clear - people who inject drugs, persons who are street-involved or low-income, or persons who are difficult-to-reach for other reasons, often experience both structural and geographic challenges to obtaining care. Community pharmacists may be the first point of contact for higher risk populations and may avoid testing and/or treatment for fear of judgement or poor treatment in hospital/specialist settings. While studies have demonstrated the feasibility of treating people receiving opioid against therapy (OAT), it remains unclear whether Canadian pharmacists can safely and effectively screen, and/or confirm HCV, work-up patients for HCV treatment, and prescribe with minimal oversight. If this model proves successful, it may have global utility especially in areas of the world where pharmacists are the initial point of contact for healthcare issues. The aim of this study is to determine whether being tested and linked care and treatment will be more effective in a community pharmacy than a referral to a tertiary care hospital for management of HCV among people on stable OAT, or other populations who experience barriers to care but use community pharmacy services.

ELIGIBILITY:
Inclusion Criteria:

1. HCV infection
2. HCV RNA > 1,000 IU/mL
3. Aged 18 to 80
4. Willingness and capacity to provide informed consent

Exclusion Criteria:

1. Presence of or history of decompensated cirrhosis. This will be defined as evidence of clinical decompensation (history of either ascites, variceal hemorrhage, or hepatic encephalopathy/confusion), and Child-Pugh-Turcotte and Model for Endstage Liver Disease (MELD) score will also be used to assess this using laboratory investigations and clinical findings.
2. Platelets < 75,000/mm3, total albumin <35 g/L, total bilirubin (total and direct) >34.2 μmol/L, International Normalized Ratio (INR) >1.5
3. History of current or past hepatocellular carcinoma
4. Hepatitis B virus (HBV) co-infection as indicated by positive testing for hepatitis B surface antigen (HBsAg +ve)or untreated HIV co-infection
5. Prior HCV antiviral therapy with direct-acting antivirals with or without peginterferon/ribavirin
6. Chronic liver disease other than mild non-alcoholic or alcoholic fatty liver disease from a cause other than HCV
7. Significant co-morbid illness that precludes inclusion in the opinion of the investigator
8. Life expectancy of less than 1 year. If clarity is required, the provider who delivered the diagnosis will be contacted.
9. Pregnancy/breast-feeding/inability to use contraception
10. Use of concomitant contraindicated drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Intention to treat by Completion Rates | 24 months
  Intention to treat direct acting antiviral (DAA) completion rates in non-cirrhotic or compensated cirrhotic patients treated with DAAs in pharmacist-led programs in community pharmacies, compared to treatment completion rates with referral and treatment in tertiary care hepatology (Toronto Centre for Liver Disease).

SECONDARY OUTCOMES:
Sustained Virologic Response by Intention-to-Treat | 24 months
  Compare Sustained Virologic Response rates by Intention to treat in both sites.
Sustained Virologic Response by modified Intention-to-Treat | 24 months
  Compare the rates of Sustained Virologic Response by modified Intention to treat (including all participants who take at least one dose of medication)
Sustained Virologic Response by Per Protocol analysis | 24 months
  Compare the rates of Sustained Virologic Response by per protocol analysis including all individuals who complete treatment in both groups.
Hepatitis C Community seroprevalence in downtown Toronto | 18 months
  Determine the seroprevalence of HCV among individuals tested in downtown Toronto.
Community Pharmacist Fibrosis Identification | 18 months
  Comparison of pharmacist-assessed fibrosis stage vs fibrosis stage assessed by hepatologist (gold standard)
Community Pharmacist Decompensation Identification | 18 months
  Comparison of pharmacist-assessed hepatic decompensation score vs hepatic decompensation assessed by hepatologist (gold standard)
Minimum Mean Time-to-Treatment | 18 months
  Determine the minimum mean time-to-treatment initiation in both groups
Community Appointment Adherence | 24 months
  Assess appointment adherence in both arms
Medication Adherence | 18 months
  Assess self-reported medication adherence at both sites
Quality of Life and Substance Use | 24 months
  Evaluate quality of life for patients with chronic liver disease (CLDQ-HCV) before and after treatment (endpoint and SV12) at both sites.
Substance Use | 24 months
  Evaluate the Maudsley Addiction Profile (MAP) before and after treatment (endpoint and SV12) at both sites.
Patient Understanding and Satisfaction | 24 months
  Compare patient understanding and satisfaction with HCV treatment with the Hepatitis Patient Satisfaction Questionnaire (HPSQ)
Reinfection | 24 months
  Assess rates of reinfection in patients who achieve Sustained Virologic Response, at 48 weeks.
Patient empowerment | 24 months
  Compare measure of patient empowerment by treatment-arm using the Health Care Empowerment (HCE) survey

CONTACTS AND LOCATIONS:
Locations (1):
- Specialty Rx Solutions, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No